CLINICAL TRIAL: NCT04264494
Title: Evaluating the Role of Intra-articular Injections of Platelet-rich Plasma (PRP) in Patients With Rheumatoid Arthritis and Its Impact on Disease Activity and Quality of Life.
Brief Title: Evaluating the Role of Intra-articular Injections of Platelet Rich Plasma (PRP) in Patients With Rheumatoid Arthritis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dalia Salah Saif (Other)
Responsible Party: Sponsor-Investigator, Dalia Salah Saif, principle investigator, Menoufia University
Organization: Menoufia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1475
Record Dates: First submitted 2020-02-03; First posted 2020-02-11 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: RA - Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): Fifty RA patients were injected intra-articularly with 3 doses of PRP in their joints
  Interventions: Procedure: PRP intra articular injection
- placebo group (Placebo Comparator): Fifty RA patients were injected intra-articularly with 3 doses of saline in their joints.
  Interventions: Procedure: NACL intra articular injection

INTERVENTIONS:
Procedure: PRP intra articular injection — Fifty RA patients were injected intra-articularly with 3 doses of PRP at 4 weeks intervals for the joints with only tenderness (arthralgia without swelling or effusion) and revaluated at 3 and 6 months post the last injection regarding the same evaluating tools.
  Other Names: PRP Injection.
  Arms: PRP group
Procedure: NACL intra articular injection — and 50 patients who serve as a control and injected intra-articularly with 3 doses of placebo (NaCl saline) at 4 weeks intervals for the joints with only tenderness (arthralgia without swelling or effusion) and revaluated at 3 and 6months post last injection regarding the same evaluating tools.
  Other Names: Placebo injection(NACL)
  Arms: placebo group

SUMMARY:
To evaluate the therapeutic effect of 3 local doses of PRP intra-articular injection in patients with RA regarding the improvement of disease activity and quality of life versus placebo.

DETAILED DESCRIPTION:
100 patients with RA fulfilling the 2010 ACR-EULAR classification criteria for RA were recruited from the outpatient clinic of the Rheumatology and Rehabilitation department. All patients were subjected to clinical and laboratory assessment, visual analog score (VAS) scale and Health Assessment Questionnaire (HAQ). Fifty patients were injected intra-articularly with 3 doses of PRP and 50 patients who serve as a control injected with 3 doses of placebo at 4 weeks intervals for the tender joints and revaluated at 1, 3 months post the last injection regarding the same evaluating tools.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as RA regarding 2010 new criteria of RA, both sex,aged20-60 years old.

Exclusion Criteria:

* Patients with Local abscess,
* systemic illness as (diabetes mellitus, malignancy),
* patients on opioids analgesics.
* pregnancy, blood disorders(coagulopathy, thrombocytopenia),

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-02-26 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale (VAS). | Change from baseline to 6 months post injection.
  the pain severity determined by the patients on scale of 0(no pain) to 10 (Agonizing pain)
Inflammatory mediators. | Change from baseline to 6 months post injection.
  By means of ELISA (IL 1 beta and TNF alpha
Health assessment questionnaire disability index. (HAQ-DI) | Change from baseline to 6 months post injection.
  Is a patient reported outcome which is usually self-administered by the patient and scales range from 0 (no difficulty) to 3 (unable to do)

SECONDARY OUTCOMES:
Disease Activity Score 28(DAS28) | At baseline,3 and 6 months post injection.
  to asses disease activity by measuring the number of tender and swollen joints,patient global assessment and ESR. values range from 2.0 (remission) to 10.0 (higher disease activity).

CONTACTS AND LOCATIONS:
Locations (1):
- Dalia Saif, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
To evaluate the therapeutic effect of 3 local doses of PRP intra-articular injection in patients with RA regarding the improvement of disease activity and quality of life versus placebo